CLINICAL TRIAL: NCT04748159
Title: Effekte Der Bauchlagerung Auf Die Vitalparameter Bei Säuglingen Mit Akuter Bronchiolitis (Masterarbeit EKNZ)
Brief Title: Effects of Prone Positioning on Vital Parameters in Infants With Acute Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Nicolas Regamey, Head of Paediatric Pulmonology, Luzerner Kantonsspital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSV Bronchiolitis
Record Dates: First submitted 2020-12-07; First posted 2021-02-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Syncytial Virus (RSV); Acute Bronchiolitis; Infant, Newborn, Disease; Infant, Premature, Diseases
Keywords: Abdominal Position; Respiratory Rate; Prone Position
MeSH Terms: conditions — Disease; Infant, Premature, Diseases | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants in prone position (Experimental): The purpose of this intervention study is to evaluate short-term effects (within one hour) of prone positioning on vital signs in infants under 12 months of age with acute RSV bronchiolitis.
  Interventions: Other: Prone position/ Abdominal position

INTERVENTIONS:
Other: Prone position/ Abdominal position — Standardized positioning of the infant in the prone position respectively abdominal position. Depending on age and size, one or two rolled towels are placed lengthwise under the baby. Both arms are placed cranially in U-position towards the head. Since the position of the head has no significant influence on lung ventilation, the head is placed according to the infant's tolerance.

SUMMARY:
This intervention study is designed to evaluate short-term effects (within one hour) of prone position on vital signs in infants under 12 months of age with acute RSV bronchiolitis. The primary objective is to investigate whether respiratory rate changes in prone position. Secondary endpoints are changes in oxygen saturation (SpO2), transcutaneous carbon dioxide partial pressure (pCO2), heart rate, and respiratory symptoms assessed by the Modified Tal Score (MTS).

DETAILED DESCRIPTION:
The study will be conducted by pediatric physical therapists (PPT). Before the start of the study, the procedure of the study as well as the recording of the measurement data in the secuTrial® database, in the Excel file and the MTS will be explained to the PPT. The ward staff will be informed about the pilot study at an early stage in order to ensure a smooth procedure parallel to the clinic activities and to initiate a physiotherapy prescription for infants with acute bronchiolitis as quickly as possible. After new registration of a physical therapy prescription of an infant, the PPT in charge will obtain informed consent from the parent or legal guardian. Each study participant will be evaluated once and preferably at the beginning of the hospitalization. If the first trial is discontinued (see discontinuation criteria), a second trial will be conducted a few hours later. Because supine positioning is promoted to prevent sudden infant death syndrome, parents are informed that prone positioning is only a measure to speed recovery from the current RSV infection and that infants are monitored throughout data collection (pulse and oxygen saturation monitors). Parents will also be informed that prone positioning should not be performed at home without monitoring.

Prior to the start of the intervention, the PPT obtain the following personal data:

* Date and time of hospital admission and physiotherapy prescription received.
* Date of birth (DD.MM. YY), age (birthday to day of intervention), sex (m/f), gestational age (gestational week), birth weight (g), ethnicity (white/other), sectio (yes/no), secondary diagnoses, positive family history (first-degree relatives) for asthma (yes/no), positive family history (first-degree relatives) for allergies (yes/no), passive smoke exposure (yes/no), breastfed (yes/no/partial), care (home, nursery, other).
* Evidence of other viruses (not tested; which virus), number of days since onset of symptoms, drug therapy, oxygen requirements, time of last feeding, type of feeding
* Date and time of onset of intervention
* Length of hospitalization (hospital admission to start of intervention)
* Position of infant when encountered prior to start of intervention (supine, lateral right, lateral left, prone, being fed, on parent's arm or lap)

If infants require oxygen administration, it is documented as high flow or low flow with the associated percent of oxygen content and liters/minute. Furthermore, the first time of oxygen administration during the hospital stay (DD.MM.YY, HH:MM), the current cycle of oxygen administration (continuous or intermittent), and the duration of oxygen administration received will be recorded. During the more than one hour of data collection, the setting of oxygen administration will not be changed by the nursing staff. The nursing staff will be informed of this prior to the start of the study.

Next, the infant's position encountered will be noted and the first data collection of vital signs (baseline, T0) will be recorded. The infant is then positioned in the prone position in a standardized manner. One to two folded towels are placed lengthwise under the infant, depending on body size. Both arms are placed cranially in a U-position towards the head. The head is placed according to any tolerance of the infant. To initially acclimate the infants to the repositioning, reassurance techniques are used by the PPT. These are individualized to the infant and involve the head, chest, and pelvis regions of the body. The calming techniques consist of gentle mobilization of the pelvis, light touching and contact breathing. The latter elicits tactile stimuli by placing the PPT's hands on various areas of the thorax and can thereby target and direct the infant's respiratory movement. After one minute, a second data collection occurs, which is labeled T1. After T1, contact with the infant is avoided by the PPT until the next measurement time points (T2 + T3). No contact is allowed to other persons during the entire data collection unless an urgent nursing or medical action is necessary due to the infant's condition (see termination criteria). After an additional 9 minutes, measurement time point T2 (T0 + 10 minutes) is collected. The last data collection occurs 60 minutes (range 45-75 minutes) after T0 and is designated T3.

If the infant turns away from the prone position, he will be repositioned to the prone position at the arrival of T1 or T2. If he turns away again after T2, T3 will not be evaluated and the trial will be terminated after T2.

Termination criteria before the start of intervention are the following conditions:

* the infant is already in the prone position. Subsequently, the infant is positioned in the supine position.
* if the infant is encountered while eating, the parents or nursing staff are instructed to position the infant in the supine position after the infant has finished eating.

In both cases, the nursing staff and the parents are then informed that the infant should not be positioned in prone position for the next few hours so that the PPT can perform the second test run a few hours later.

The following parameters are recorded in analogous order at each measurement time point, that is, T0 to T3. The primary outcome is the change in infant respiratory rate after intervention has occurred. This parameter is determined first and for a precise result by auscultation with the help of a stethoscope by the respective PPT. In this process, the breaths are counted in the period of one minute. Secondarily, the oxygen saturation SpO2(%) and heart rate (beats/minute) are measured using the pulse oximeter Philips IntelliVue MP70 Neonatal ®. Transcutaneous partial pressure of carbon dioxide (pCO2) is measured using a transcutaneous pCO2 probe on the infant's thorax and can be read on the TCM4 Series ® radiometer. In addition, evaluation is performed by Modified Tal Score (MTS) and recording of cough. If coughing occurred between T1 and T3, it is noted whether it was productive or non-productive and occurred at the momentary measurement time or between the measurement time points. The feasibility regarding the parents is recorded externally by the secuTrial® database using an Excel file. For each infant, the following is documented in the Excel file:

* Did the parents consent to study participation? Yes/ No
* Did the parents request discontinuation during data collection? Yes/ No
* Did the parents independently terminate the intervention by their own actions (e.g., by picking up the infant)? Yes/ No
* Other incidents can be noted in free text

Termination criteria: Prone positioning is terminated if the SpO2 value drops below 80% over a period of 15 seconds or below 85% over a period of one minute. Other discontinuation criteria include vomiting, massive coughing fit, apnea, incessant crying, turning away from the prone position after T2, and discontinuation after parental request. If abortion from the prone position is necessary, depending on the PPT's time availability, another attempt at data collection will be made a few hours later. If the second test run is aborted, time "T" and reason for abortion will be documented. If discontinuation of both intervention runs was necessary, the first test run will be included in the data analysis. Nevertheless, the results of both intervention runs are saved so that any subsequent analyses can be performed.

ELIGIBILITY:
Inclusion Criteria:

* Infants hospitalized due to RSV at the Lucerne Children's Hospital in the 2020 RSV season
* Infants under twelve months with a mild to moderate severity of acute bronchiolitis
* positive RSV Test: rapid antigen test or detection of nucleic acids by PCR in nasopharyngeal secretion

Exclusion Criteria:

* Infants who are in a life-threatening condition and require intensive care

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change of the respiratory rate at 45-75 minutes | Time 3 = Change from baseline at 45-75 minutes.
  This parameter is determined first and by visual observation of the respective PPT. The breaths are counted in a period of one minute.

SECONDARY OUTCOMES:
Respiratory rate: Baseline | Time 0 = Collection of measurement data for the baseline. Repositioning of the child in prone position.
  This parameter is determined first and by visual observation of the respective PPT. The breaths are counted in a period of one minute.
Change of the respiratory rate at 1 minute | Time 1 = Change from baseline at 1 minute.
  This parameter is determined first and by visual observation of the respective PPT. The breaths are counted in a period of one minute.
Change of the respiratory rate at 10 minutes | Time 2 = Change from baseline at 10 minutes.
  This parameter is determined first and by visual observation of the respective PPT. The breaths are counted in a period of one minute.
Oxygen saturation (SpO2): Baseline | Time 0: Collection of measurement data for the baseline. Repositioning of the child in prone position.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Change of oxygen saturation at 1 minute | Time 1 = Change from baseline at 1 minute.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Change of oxygen saturation at 10 minutes | Time 2 = Change from baseline at 10 minutes.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Change of oxygen saturation at 45-75 minutes | Time 3 = Change from baseline at 45-75 minutes.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Transcutaneous carbon dioxide partial pressure (pCO2): Baseline | Time 0: Collection of measurement data for the baseline. Repositioning of the child in prone position.
  Is performed with a transcutaneous pCO2 probe on the thorax of the infant and can be read on the radiometer TCM4 Series ®.
Change of transcutaneous carbon dioxide partial pressure at 1 minute | Time 1 = Change from baseline at 1 minute.
  Is performed with a transcutaneous pCO2 probe on the thorax of the infant and can be read on the radiometer TCM4 Series ®.
Change of transcutaneous carbon dioxide partial pressure at 10 minutes | Time 2 = Change from baseline at 10 minutes.
  Is performed with a transcutaneous pCO2 probe on the thorax of the infant and can be read on the radiometer TCM4 Series ®.
Change of transcutaneous carbon dioxide partial pressure at 45-75 minutes | Time 3 = Change from baseline at 45-75 minutes.
  Is performed with a transcutaneous pCO2 probe on the thorax of the infant and can be read on the radiometer TCM4 Series ®.
Heart rate: Baseline | Time 0: Collection of measurement data for the baseline. Repositioning of the child in prone position.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Change of the heart rate at 1 minute | Time 1 = Change from baseline at 1 minute.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Change of the heart rate at 10 minutes | Time 2 = Change from baseline at 10 minutes.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Change of the heart rate at 45-75 minutes | Time 3 = Change from baseline at 45-75 minutes.
  Measurement using the Philips IntelliVue MP70 Neonatal ® pulse oximeter.
Symptom-Score - Modified Tal Score (MTS): Baseline | Time 0: Collection of measurement data for the baseline. Repositioning of the child in prone position.
  Calculation of the Modified Tal Score (MTS). Minimum value: 0. Maximum value: 12. A higher value of MTS indicates more severe symptoms of affected RSV bronchiolitis infants.
Symptom-Score - MTS at 1 minute | Time 1 = Change from baseline at 1 minute.
  Calculation of the Modified Tal Score (MTS). Minimum value: 0. Maximum value: 12. A higher value of MTS indicates more severe symptoms of affected RSV bronchiolitis infants.
Symptom-Score MTS at 10 minutes | Time 2 = Change from baseline at 10 minutes.
  Calculation of the Modified Tal Score (MTS). Minimum value: 0. Maximum value: 12. A higher value of MTS indicates more severe symptoms of affected RSV bronchiolitis infants.
Symptom-Score: MTS | Time 3 = Change from baseline at 45-75 minutes.
  Calculation of the Modified Tal Score (MTS). Minimum value: 0. Maximum value: 12. A higher value of MTS indicates more severe symptoms of affected RSV bronchiolitis infants.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Regamey, MD, Principal Investigator — Luzerner Kinderspital
Locations (1):
- Kinderspital Luzern, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No